CLINICAL TRIAL: NCT02070120
Title: CALIBER - A Phase II Randomised Feasibility Study of Chemoresection and Surgical Management in Low Risk Non Muscle Invasive Bladder Cancer
Brief Title: Investigating Bladder Chemotherapy Instead of Surgery for Low Risk Bladder Cancer
Acronym: CALIBER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2013/10041; 2013-005095-18 (EudraCT Number)
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Bladder Cancer
Keywords: Nonmuscle invasive bladder cancer (NMIBC); Mitomycin C; Chemoresection
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoresection (Experimental): 4 once weekly outpatient intravesical instillations 40mg Mitomycin C
  Interventions: Drug: Mitomycin C
- Surgical Management (Other): Surgical management according to local practice
  Interventions: Procedure: Surgical Management

INTERVENTIONS:
Drug: Mitomycin C — Patients assigned to the chemoresection group will receive 4 once weekly intravesical instillations of 40mg MMC as outpatients.
  Other Names: MMC
  Arms: Chemoresection
Procedure: Surgical Management — Patients in this group should be treated according to local practice. Surgical interventions may include transurethral resection (TUR) or ablation.
  Arms: Surgical Management

SUMMARY:
Patients diagnosed with low risk non-muscle invasive bladder cancer (NMIBC) are at risk of frequent low grade recurrence, which usually necessitates surgical intervention under general anaesthetic. This multicentre study aims to establish the short term efficacy of chemoresection using chemotherapy within the bladder for the treatment of NMIBC.

Should the levels of complete response following chemoresection meet predefined criteria, a larger phase III trial would be developed to assess longer term disease related endpoints, with the aim of standardising management of recurrent low risk NMIBC and potentially removing the need for over a thousand patients each year to undergo surgery.

DETAILED DESCRIPTION:
CALIBER is a two stage phase II, multicentre, randomised controlled trial (RCT). A control group has been included to provide prospective data about surgical management and outcomes and assess feasibility of recruitment to a randomised study.

Stage 1: 80 patients will be recruited with treatment allocated 2:1 by randomisation between chemoresection and surgical management.

Stage 2: If the stop/go activity criteria at the end of stage 1 indicate that recruitment should continue, 9 additional participants will be recruited, all of whom will receive chemoresection.

Patients assigned to the chemoresection group will receive 4 once weekly intravesical instillations of 40mg Mitomycin C (MMC) as outpatients. This treatment will be delivered via catheter under local anaesthetic.

Patients assigned to the surgical management group will receive the standard surgical management in use at their hospital for treatment of recurrence which may include a single post-operative installation of 40mg MMC within 24 hours.

All participants will be followed up at 3 weeks from the start of treatment (ie at time of final MMC instillation for chemoresection group) and each will receive a cystoscopy three months from the end of treatment to assess response, in accordance with European Association of Urology (EAU) guidelines.

Subsequent cystoscopic follow up will take place 12 months after treatment if recurrence-free at 3 months and then annually.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* NMIBC recurrence following original diagnosis of low risk NMIBC (defined as Ta G1 or Ta G2 (Ta low grade) with a risk of recurrence score of ≤6 using EORTC risk tables
* Histologically confirmed Transitional-cell carcinoma (TCC) at original diagnosis
* Aged 16 or over
* Satisfactory pre-treatment haematology values and serum creatinine < 1.5 x Upper Limit of Normal (ULN)
* Negative pregnancy test for women of child-bearing potential

Exclusion Criteria:

* Any history of: grade 3/high grade or ≥T1 transitional cell carcinoma, concomitant carcinoma in situ, more than 7 tumours at one diagnosis or more than 1 recurrence per year since initial diagnosis or in the past five years, whichever is shorter
* Any history of histologically confirmed non-TCC bladder cancer
* Trial entry recurrence identified within 11.5 months of the date of the original diagnosis
* Any prior treatment of the trial entry recurrence (including biopsy)
* Previous MMC chemotherapy other than a single instillation at diagnostic surgery
* Known allergy to MMC
* Carcinoma involving the prostatic urethra or upper urinary tract (participants should have had imaging of the upper urinary tract within 2 years prior to randomisation)
* Known or suspected reduced bladder capacity (<100ml)
* Significant bleeding disorder
* Female patients who are breast-feeding or are of childbearing potential and unwilling or unable to use adequate non-hormonal contraception. Male patients should also use contraception if sexually active.
* Active or intractable urinary tract infection
* Urethral stricture or anything impeding the insertion of a catheter
* Large narrow neck diverticula
* Significant urinary incontinence
* Any other conditions that in the Principal Investigator's opinion would contraindicate protocol treatment
* Unable or unwilling to comply with study procedures or follow up schedule

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Complete response rate with chemoresection | 3 months
  Defined as an absence of any tumour following chemoresection and will be assessed visually at 3 month check cystoscopy by patients' urologists. A biopsy of the tumour bed would take place to confirm visual assessment of complete response.

SECONDARY OUTCOMES:
Treatment compliance in chemoresection group | Duration of treatment (3 weeks)
  Patients who receive 4 MMC instillations with no more than 14 days between each instillation will be described as fully compliant.
Salvage surgery rates | 3 years
  Assessing trans-urethral resection and biopsy rates following initial treatment in both treatment groups
Progression-free survival | 3 years
  Defined as time from randomisation to the first of muscle invasive bladder recurrence, recurrence in the pelvic nodes, distant metastatic recurrence or death from any cause.
Toxicity (NCI Common Toxicity Criteria for Adverse Effects (CTCAE) V4 and Clavien Dindo grade (in surgical group)) | up to 12 months
  Measuring side effects of both treatments using clinician reported toxicity scales
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) and Superficial Bladder Cancer (BLS24) questionnaire | up to 12 months
  Assessing side effects and impact of both treatments on patient reported quality of life.
Health service utilisation | up to 12 months
  Assessed using prospective data collection of health resource usage.
Recurrence free interval | up to 12 months
  Time from end of treatment to first relapse, in patients confirmed recurrence free at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Mostafid, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (38):
- United Kingdom (38):
  - Macclesfield District General Hospital, Macclesfield, Cheshire
  - James Cook University Hospital, Middlesbrough, Cleveland
  - West Cumberland Hospital, Whitehaven, Cumbria
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Derriford Hospital, Plymouth, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Dorset County Hospital, Dorchester, Dorset
  - Cumberland Infirmary, Carlisle, England
  - Broomfield Hospital, Chelmsford, Essex
  - Princess Alexandra Hospital, Harlow, Essex
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Gloucestershire Royal Hospital, Gloucester, Gloucestershire
  - Royal Oldham Hospital, Manchester, Greater Manchester
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Southampton General Hospital, Southampton, Hampshire
  - Hereford County Hospital, Hereford, Herefordshire
  - Darent Valley Hospital, Dartford, Kent
  - Medway Maritime Hospital, Gillingham, Kent
  - Royal Preston Hospital, Preston, Lancashire
  - Leicester General Hospital, Leicester, Leicestershire
  - Northwick Park Hospital, Harrow, Middlesex
  - Churchill Hospital, Headington, Oxfordshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Ipswich Hospital, Ipswich, Suffolk
  - Croydon University Hospital, Croydon, Surrey
  - Royal Surrey County Hospital, Guildford, Surrey
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - New Cross Hospital, Wolverhampton, West Midlands
  - St Richard's Hospital, Chichester, West Sussex
  - Worthing Hospital, Worthing, West Sussex
  - Pinderfields General Hospital, Wakefield, West Yorkshire
  - Kidderminster Hospital, Kidderminster, Worcestershire
  - Alexandra Hospital, Redditch, Worcestershire
  - Worcester Royal Hospital, Worcester, Worcestershire
  - St James's University Hospital, Leeds, Yorkshire
  - University College Hospital, London
  - Withington Hospital, Manchester
  - Wythenshawe Hospital, Manchester

REFERENCES:
- [Result] Mostafid AH, Porta N, Cresswell J, Griffiths TRL, Kelly JD, Penegar SR, Davenport K, McGrath JS, Campain N, Cooke P, Masood S, Knowles MA, Feber A, Knight A, Catto JWF, Lewis R, Hall E. CALIBER: a phase II randomized feasibility trial of chemoablation with mitomycin-C vs surgical management in low-risk non-muscle-invasive bladder cancer. BJU Int. 2020 Jun;125(6):817-826. doi: 10.1111/bju.15038. Epub 2020 Apr 3. PMID 32124514